CLINICAL TRIAL: NCT04770961
Title: Erector Spinae Plane Block for Minimally Invasive Mitral Surgery
Brief Title: Erector Spinae Plane Block for Minimally Invasive Mitral Valve Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-29298
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Mitral Regurgitation; Mitral Valve Insufficiency; Mitral Valve Prolapse
Keywords: mitral valve replacement; mitral valve repair; mitral valve surgery; erector spinae plane; minimally invasive surgery
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Prolapse | interventions — Ropivacaine; Sodium Chloride; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoablation (Sham Comparator): 1. Cryoablation of intercostal nerves + Sham ESP catheter with saline infusion.
  Interventions: Procedure: Erector spinae plane catheter with saline
- ESP + Cryoablation (Experimental): 2. Cryoablation of intercostal nerves + ESP catheter with local anesthetic infusion.
  Interventions: Procedure: Erector spinae plane catheter with 0.5% Ropivacaine

INTERVENTIONS:
Procedure: Erector spinae plane catheter with 0.5% Ropivacaine — Ultrasound guided, right sided, ESP catheter inserted at the level of T5. 20 cc injection of 0.5% Ropivacaine is injected at the time of catheter placement. Postoperatively, a programmed intermittent bolus infusion of 0.2% Ropivacaine will be delivered via the ESP catheter.
  Arms: ESP + Cryoablation
Procedure: Erector spinae plane catheter with saline — Ultrasound guided, right sided, ESP catheter inserted at the level of T5. 20 cc injection of saline is injected at the time of catheter placement. Postoperatively, a programmed intermittent bolus infusion of saline will be delivered via the ESP catheter.
  Other Names: Sham
  Arms: Cryoablation

SUMMARY:
The goal of this project is to study whether local anesthetic via the erector spinae plane (ESP) block may be beneficial in minimally invasive mitral valve surgery (MIMVS).

DETAILED DESCRIPTION:
This is a double blinded randomized controlled trial comparing a control group receiving cryoablation and sham block with an intervention group receiving cryoablation and ESP catheter. The primary outcome is total oral morphine equivalent (OME) consumption within the first 48 hours of recovery including intra-operative usage. Secondary outcomes to be evaluated would include pain scores, functional milestones like time to extubation, time to first PO intake, time to ambulation, time to chest tube removal, length of ICU and total hospital stay, complications, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Elective mitral valve repair or replacement
* Planned minimally invasive approach

Exclusion Criteria:

* Non-English speaking
* Emergency surgery
* Planned or unplanned sternotomy
* Previous history of sternotomy and cardiac surgery
* Allergy to ropivacaine
* Patients taking more than 60 OMEs per day
* Patients with coagulopathy or taking anticoagulant with laboratory findings contraindicated for ESP catheter

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Total opiate consumption | 48 hours.
  Total oral morphine equivalent (milligram) consumption within the first 48 hours of recovery including intra-operative usage, extracted from electronic medical record.

SECONDARY OUTCOMES:
Pain score | 48 hours
  Pain Scores will be measured on the Visual Analog Scale (VAS), the score ranges from 0-10, zero indicating no pain and 10 indicating the worst pain, assessed by nursing staff, and extracted from electronic medical record.
Time to extubation. | Within 30 days from end of operation.
  Length from ICU arrival to endotracheal extubation (minutes). If extubated in the operating room, the time will be 0 minute. Extracted from electronic medical record.
Time to first oral intake | Within 30 days from end of operation.
  Length from ICU arrival to the time of first oral intake (hours). Extracted from electronic medical record.
Time to ambulation | Within 30 days from end of operation.
  Length from ICU arrival to the time of first ambulation (hours). Extracted from electronic medical record.
Time to chest tube removal | Within 30 days from end of operation.
  Length from ICU arrival to the time of last chest tube removal (hours). Extracted from electronic medical record.
Length of intensive care stay | Within 30 days from end of operation.
  Length from ICU arrival to ICU discharge (hours). Extracted from electronic medical record.
Length of hospital stay | Within 30 days from end of operation.
  Length from ICU arrival to hospital discharge (Hours). Extracted from electronic medical record.
Patient self-reported experience with surgery and postoperative recovery | 30 days after hospital discharge.
  Based on questionnaires regarding the patient's experience with the efficacy of pain control and the satisfaction with postoperative recovery with scores from 1 (not satisfied at all) to 5 (very satisfied) conducted over telephone or video conferencing.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Cui, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No